CLINICAL TRIAL: NCT02243267
Title: Biospecimens for the Diagnosis, Treatment and Prevention of Colorectal Cancer
Brief Title: GI SPORE Colon Biosample Protocol
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Missy Tuck, Project manager, University of Michigan
Other Study IDs: HUM00064405
Record Dates: First submitted 2014-09-11; First posted 2014-09-17 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: Colon Cancer Colon Cancer Prevention
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Plasma Buffy Coat Tissue Stool Urine
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: sample collection

SUMMARY:
The investigators are creating a data and specimen repository to study causes , early detection, prevention and treatment of colon and rectal cancer. The investigators are collecting data and specimens (blood, stool, urine and tissue) from people who have colon or rectal cancer, or who are risk for developing colorectal cancer or had normal colonoscopies. Data and samples are held in the repository until there are enough to be used for a large study or until there are new techniques that can be used to test them. The GI SPORE Program at the University of Michigan maintains a repository of specimens for colorectal diseases that the investigators hope will help fuel new research. The investigators hope that this work may lead to new treatments or earlier detection of colorectal cancer or improved diagnosis and treatment of other colon and rectal diseases.

ELIGIBILITY:
Inclusion Criteria:

5.2 General Eligibility Criteria 5.2.1 Overall Inclusion

1. Adults 18 years of age or older
2. Willing to sign informed consent.
3. Able to tolerate removal of up to 50 ml of blood

5.2.2 Overall Exclusion Criteria

1. Pregnant, lactating
2. Unable to understand English
3. Known HIV/AIDS or Hepatitis C

5.3 Disease or Control Specific Eligibility Criteria 5.3.1 Unaffected Healthy Individuals (Healthy Controls)

1. No prior colorectal neoplasia
2. Undergoing colonoscopy in the next 3-4 months OR had an endoscopically normal colonoscopy within the previous 6 months.
3. Not prepped for colonoscopy at the time of blood draw
4. No personal history of colorectal cancer
5. No personal history of other cancers in the last 5 years (except basal/squamous skin lesions)

5.3.2 Prior non-invasive colorectal neoplasia (Adenoma surveillance)

1. Personal history of one or more adenomas or sessile serrated polyps in colon
2. Undergoing colonoscopy in the next 3-4 months
3. Not prepped for colonoscopy at the time of blood draw
4. No personal history of colorectal cancer
5. No personal history of other cancers in the last 5 years (except basal/squamous skin lesions)

5.3.3 New Diagnosis of Colon Adenocarcinoma (untreated, new colon CA)

1. Newly diagnosed colon adenocarcinoma, any stage
2. No treatment received yet
3. Not prepped for colonoscopy or surgery at the time of blood draw

5.3.4 New Diagnosis of Rectal Adenocarcinoma (untreated, new rectal CA)

1. Newly diagnosed rectal adenocarcinoma, any stage
2. No treatment received yet
3. Not prepped for colonoscopy or surgery at the time of blood draw

5.3.5 Colorectal Cancer (less than 5 years ago) (current/recent CRC)

1. Personal history of colorectal adenocarcinoma within the last 5 years
2. Not prepped for colonoscopy at the time of blood draw
3. No personal history of other cancers in the last 5 years (except basal/squamous skin lesions)

5.3.6 Colorectal Cancer (greater than 5 years ago)(remote history of colorectal cancer)

1. Personal history of colorectal adenocarcinoma greater than 5 years ago
2. Not prepped for colonoscopy at the time of blood draw

5.3.7 Hereditary Cancer syndrome (confirmed or suspected) (genetic risk of colorectal cancer)

1. Personal or family history which meets clinical criteria for genetic evaluation for a hereditary cancer syndrome
2. Not prepped for colonoscopy at the time of blood draw

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of the University of Michigan Health System
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2014-09; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
New Biomarker for colon cancer detection | 6 years
  To create a longitudinal biorepository from individuals with colorectal cancer, those who are high risk for developing colorectal cancer, and screened, endoscopically normal controls including a reference set of well annotated, pathologically confirmed tissue, plasma, serum, and white blood cell biosamples and corresponding demographic, risk, and clinical treatment data for improved colon cancer detection.
Response to Treatment | 6 years
  To create a longitudinal biorepository from individuals with colorectal cancer, those who are high risk for developing colorectal cancer, and screened, endoscopically normal controls including a reference set of well annotated, pathologically confirmed tissue, plasma, serum, and white blood cell biosamples and corresponding demographic, risk, and clinical treatment data for improved colon cancer detection.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States